CLINICAL TRIAL: NCT00778895
Title: Clinical Study in Children, 6 Months to 3 Years of Age, to Assess the Immunogenicity and Safety of Two Dose Levels of Thimerosal-free Fluviral® Vaccine, Using a Licensed Influenza Virus Vaccine, Vaxigrip® as the Control
Brief Title: Clinical Study in Children, 6 Months to 3 Years of Age, to Assess Two Dose Levels of an Experimental Flu Vaccine, Using a Licensed Influenza Virus Vaccine, Vaxigrip® as the Control
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 111635
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Results first posted 2013-07-09 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2016-10

CONDITIONS: Influenza
Keywords: Flu; Safety; Immunogenicity; Flu vaccine; Influenza; Virus
MeSH Terms: conditions — Influenza, Human; Virus Diseases | interventions — Influenza Vaccines; vaxigrip

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Fluviral F1 Group (Experimental): Subjects 6 months to 3 years of age received if primed, 1 dose of formulation 1 of Fluviral vaccine at Day 0 and if unprimed, 2 doses of formulation 1 of Fluviral vaccine at Day 0 and approximately Day 28. The vaccine was administered intramuscularly in the anterolateral part of the thigh (if the subject was less than 12 months) or in the deltoid region of the arm.
  Interventions: Biological: GSK Biologicals' influenza vaccine GSK1557482A
- Fluviral F2 Group (Experimental): Subjects 6 months to 3 years of age received if primed, 1 dose of formulation 2 of Fluviral vaccine at Day 0 and if unprimed, 2 doses of formulation 1 of Fluviral vaccine at Day 0 and approximately Day 28. The vaccine was administered intramuscularly in the anterolateral part of the thigh (if the subject was less than 12 months) or in the deltoid region of the arm.
  Interventions: Biological: GSK Biologicals' influenza vaccine GSK1557482A
- Vaxigrip Group (Active Comparator): Subjects 6 months to 3 years of age received if primed, 1 dose of Vaxigrip vaccine at Day 0 and if unprimed, 2 doses of Vaxigrip vaccine at Day 0 and approximately Day 28. The vaccine was administered intramuscularly in the anterolateral part of the thigh (if the subject was less than 12 months) or in the deltoid region of the arm.
  Interventions: Biological: Vaxigrip

INTERVENTIONS:
Biological: GSK Biologicals' influenza vaccine GSK1557482A — one IM injection at Day 0 for primed subjects (defined as subjects who had a prior 2-dose priming influenza immunization) or two IM injections at Day 0 and approximately Day 28 for un-primed subjects (defined as subjects who have not previously received a complete 2-dose priming influenza immunization).
  Other Names: Fluviral
  Arms: Fluviral F1 Group; Fluviral F2 Group
Biological: Vaxigrip — one IM injection at Day 0 for primed subjects (defined as subjects who had a prior 2-dose priming influenza immunization) or two IM injections at Day 0 and approximately Day 28 for un-primed subjects (defined as subjects who have not previously received a complete 2-dose priming influenza immunization).
  Arms: Vaxigrip Group

SUMMARY:
Children younger than 5 years of age are at high risk for severe influenza disease (flu) and hospitalization due to flu. Scientists are in the process of re-evaluating the dosing initially based on whole virus vaccines to improve their efficacy in infants. In this study, we will compare two different dose levels of GSK1557482A flu vaccine. Another already approved flu vaccine made by a different company will be used as a control.

DETAILED DESCRIPTION:
This is a study of two different dose levels of a new formulation of flu vaccine for the 2008/2009 flu season using the World Health Organization recommended virus strains. Subjects will be randomly put into one of three different groups to receive either one or two doses of:

0.25 mL dose of the new flu vaccine, or 0.5 mL dose of the new flu vaccine or the licensed Vaxigrip flu vaccine (control) The parents of the subjects and the study doctor and nurses will not know the group of their child until the study is completed.

The children will be vaccinated with either one dose or two doses depending on whether or not they have received a flu vaccine before. The doctor will decide on the schedule for each child based on the information provided by the parents. The active phase of the study will last approximately two months for children receiving two doses and one month for those receiving a single dose. An extended safety follow-up will continue until Study Month 6.

Two blood samples will be taken from each subject. These will be used to evaluate how well the vaccine works in the children and which dose level works best compared to the control.

The parents will fill in a diary card for four days to record any reactions or symptoms which may occur after vaccination. Parents will also keep a record of other symptoms that may occur between vaccinations and up to six months after the first vaccination and will keep a record of any medication their child takes in this time period.

ELIGIBILITY:
Inclusion Criteria:

* A male or female child 6 months to < 3 years of age at the time of the vaccination, regardless of previous administration of influenza vaccine in a previous season;
* Subjects must be in good health established by medical history and physical examination before entering into the study;
* Subjects having a parent/guardian who the investigator believes can and will comply with the requirements of the protocol should be enrolled in the study;
* Written informed consent obtained from the subject's parent/guardian.
* Parents/guardian access to a consistent means of telephone contact, land line or mobile

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the administration of the study vaccine or planned use during the study period. Routine, registered childhood vaccinations are not an exclusion criterion;
* History of hypersensitivity to any vaccine;
* History of allergy to or reactions likely to be exacerbated by, any component of the vaccine including egg, chicken protein, formaldehyde, or sodium deoxycholate;
* History of any congenital, acquired, or iatrogenic immunodeficiency state (current or potential) including HIV infection, disorders of the lymphoid system or bone marrow, or chronic administration (defined as more than 14 consecutive days) of immunosuppressant or other immune-modifying drugs within 3 months prior to the administration of the study vaccine.
* Acute disease at the time of enrolment.
* History of Guillain Barré syndrome within 6 weeks of receipt of prior inactivated influenza virus vaccine;
* Any significant disorder of blood coagulation or treatment with vitamin K antagonists; or any known disorder of hemostasis;
* Receipt of any immunoglobulins and/or any blood products within three months of study enrollment or planned administration of any of these products during the study period.
* Receipt of a non-study related influenza vaccine outside of this study and during the current (2008-09) influenza immunization campaign.
* Any use of analgesics/antipyretics 12 hours before receipt of vaccine.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 390 (Actual)
Dates: Start 2008-11-10; Primary Completion 2009-08-19 (Actual); Study Completion 2009-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- Canada (17):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Langley, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Mount Pearl, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Newmarket, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Charlottetown, Prince Edward Island
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Ste-Foy, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Langley JM, Vanderkooi OG, Garfield HA, Hebert J, Chandrasekaran V, Jain VK, Fries L. Immunogenicity and Safety of 2 Dose Levels of a Thimerosal-Free Trivalent Seasonal Influenza Vaccine in Children Aged 6-35 Months: A Randomized, Controlled Trial. J Pediatric Infect Dis Soc. 2012 Mar;1(1):55-63. doi: 10.1093/jpids/pis012. Epub 2012 Mar 1. PMID 23687572
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 111635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111635 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were differentiated according to priming status. Primed Subjects - subjects who had a prior 2-dose priming influenza immunization received a 1-dose vaccination course in the study. Unprimed Subjects - subjects who had not previously received a complete 2-dose priming influenza immunization received a 2-dose vaccination course in the study.
Pre-assignment Details: Study comprised an Active phase of approximately 2 months and a post-vaccination 180 day extended safety follow-up period (ESFU phase).
  374 subjects out of the 390 who were enrolled in the study were vaccinated. Remaining subjects were not included in the participant flow as started as they failed to meet protocol criteria.
Period: Active Phase
Arm/Group | Fluviral F1 Group | Fluviral F2 Group | Vaxigrip Group
Started | 164 | 167 | 43
Completed | 157 | 161 | 43
Not Completed | 7 | 6 | 0
Not completed — Adverse Event | 3 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Other | 2 | 0 | 0
Period: ESFU Phase
Arm/Group | Fluviral F1 Group | Fluviral F2 Group | Vaxigrip Group
Started | 164 | 167 | 43
Completed | 153 | 155 | 41
Not Completed | 11 | 12 | 2
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 0
Not completed — Lost to Follow-up | 6 | 7 | 2
Not completed — Other | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluviral F1 Group | Fluviral F2 Group | Vaxigrip Group | Total
Number analyzed (Participants) | 164 | 167 | 43 | 374
Age, Continuous [Mean (Standard Deviation); unit: Years] | 18.2 (9.06) | 17.5 (8.27) | 17.0 (8.33) | 17.7 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 83 | 26 | 179
  Male | 94 | 84 | 17 | 195

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms After Vaccination
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any solicited local symptom reported regardless of intensity grade. Grade 3 pain = Cried when limb was moved/spontaneously painful. Grade 3 redness and swelling were defined as redness/swelling above 50 millimeters (mm). This primary outcome measure was assessed for Fluviral F1 Group and Fluviral F2 Group respectively as per the study protocol.
Time Frame: During the 4-day follow-up period (Days 0-3) after any vaccination
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with at least one vaccine administration documented and symptom sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluviral F1 Group | Fluviral F2 Group
Number analyzed (Participants) | 161 | 164
Participants
  Any pain | 45 | 55
  Grade 3 pain | 1 | 1
  Any redness | 49 | 54
  Grade 3 redness | 0 | 0
  Any swelling | 22 | 24
  Grade 3 swelling | 0 | 0

2. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms After Vaccination
Description: Symptoms assessed were drowsiness, irritability, loss of appetite and fever. Any was defined as occurrence of any general symptom regardless of their intensity grade or relationship to vaccination. Any fever = Axillary temperature ≥ 38.0 degrees Celsius (°C). Grade 3 fever = Axillary temperature ≥ 39.0°C. For other symptoms, grade 3 was defined as an adverse event which prevented normal everyday activities. Related = A general symptom assessed by the investigator as causally related to vaccination. This primary outcome measure was assessed for Fluviral F1 Group and Fluviral F2 Group respectively as per the study protocol.
Time Frame: During the 4-day follow-up period (Days 0-3) after any vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluviral F1 Group | Fluviral F2 Group
Number analyzed (Participants) | 161 | 163
Participants
  Any drowsiness | 54 | 65
  Grade 3 drowsiness | 3 | 3
  Related drowsiness | 44 | 52
  Any irritability | 81 | 83
  Grade 3 irritability | 9 | 7
  Related irritability | 62 | 69
  Any loss of appetite | 50 | 54
  Grade 3 loss of appetite | 5 | 5
  Related loss of appetite | 37 | 43
  Any fever | 16 | 9
  Grade 3 fever | 4 | 1
  Related fever | 10 | 6

3. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs) After Vaccination
Description: Unsolicited AEs covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = Occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Grade 3 = Occurrence of any unsolicited AE that prevented normal, everyday activities. Related = Occurrence of an unsolicited AE assessed by the investigator to be causally related to study vaccination. This primary outcome measure was assessed for Fluviral F1 Group and Fluviral F2 Group respectively as per the study protocol.
Time Frame: During the 28-day follow-up period (Days 0-27) after vaccination
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluviral F1 Group | Fluviral F2 Group
Number analyzed (Participants) | 164 | 167
Participants
  Any unsolicited AE(s) | 108 | 112
  Grade 3 unsolicited AE(s) | 19 | 17
  Related unsolicited AE(s) | 26 | 30

4. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Medically-attended Adverse Events (MAEs) After Vaccination
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any MAE(s) = Occurrence of any MAE(s) regardless of intensity grade or relation to vaccination.
  Analysis of intensity and relationship to vaccination of MAEs was not performed.
  This primary outcome measure was assessed for Fluviral F1 Group and Fluviral F2 Group respectively as per the study protocol.
Time Frame: During the 28-day post-vaccination period
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Fluviral F1 Group | Fluviral F2 Group
Number analyzed (Participants) | 164 | 167
Participants | 52 | 40

5. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Medically-attended Adverse Events (MAEs) After Vaccination
Description: as for outcome 4
Time Frame: During the 6-month safety follow up after vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Fluviral F1 Group | Fluviral F2 Group
Number analyzed (Participants) | 164 | 167
Participants | 73 | 57

6. Primary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs) After Vaccination
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any SAE(s) = Occurrence of any SAE(s) regardless of intensity grade or relation to vaccination. Related SAE(s) = Occurrence of any SAE(s) assessed by the investigator as causally related to vaccination.
  This primary outcome measure was assessed for Fluviral F1 Group and Fluviral F2 Group respectively as per the study protocol.
Time Frame: During the 28-day post-vaccination period
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Fluviral F1 Group | Fluviral F2 Group
Number analyzed (Participants) | 164 | 167
Participants
  Any SAE(s) | 1 | 1
  Related SAE(s) | 0 | 0

7. Primary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs) After Vaccination
Description: as for outcome 6
Time Frame: During the 6-month safety follow up after vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Fluviral F1 Group | Fluviral F2 Group
Number analyzed (Participants) | 164 | 167
Participants
  Any SAE(s) | 1 | 1
  Related SAE(s) | 0 | 0

8. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies
Description: Titers are presented as geometric mean titers (GMTs). The reference cut-off value was the seropositivity cut-off of 1:10. Antibodies assessed were antibodies against the A/Brisbane (H1N1), A/Uruguay (H3N2) and B/Florida flu strains.
Time Frame: At Day 0 [PRE] and at Day 28 (for primed subjects) and Day 56 (for unprimed subjects) [POST]
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity which included all vaccinated and eligible subjects for whom data concerning immunogenicity outcome measures were available and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluviral F1 Group | Fluviral F2 Group | Vaxigrip Group
Number analyzed (Participants) | 131 | 132 | 36
Titer
  A/Brisbane (H1N1) strain [PRE] | 8.3 [6.9 to 10.1] | 8.5 [7.0 to 10.3] | 8.1 [5.9 to 11.0]
  A/Brisbane (H1N1) strain [POST] | 56.3 [39.5 to 80.2] | 70.7 [50.7 to 98.6] | 120.9 [73.4 to 199.0]
  A/Uruguay (H3N2) strain [PRE] | 7.0 [5.9 to 8.3] | 9.2 [7.4 to 11.4] | 7.3 [4.9 to 11.1]
  A/Uruguay (H3N2) strain [POST] | 64.5 [48.2 to 86.4] | 89.5 [67.4 to 119.0] | 97.8 [59.0 to 162.4]
  B/Florida strain [PRE] | 7.9 [6.7 to 9.4] | 7.9 [6.6 to 9.4] | 10.8 [6.9 to 16.9]
  B/Florida strain [POST] | 128.7 [100.3 to 165.1] | 163.7 [130.1 to 206.0] | 190.3 [119.0 to 304.3]

9. Secondary Outcome: Number of Subjects Seroconverted to HI Antibodies
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥1:40, or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The flu strains assessed were the A/Brisbane (H1N1), A/Uruguay (H3N2) and B/Florida.
Time Frame: At Day 28 (for primed subjects) and at Day 56 (for unprimed subjects) [POST]
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Fluviral F1 Group | Fluviral F2 Group | Vaxigrip Group
Number analyzed (Participants) | 131 | 132 | 36
Participants
  A/Brisbane (H1N1) [POST] | 67 | 82 | 29
  A/Uruguay (H3N2) [POST] | 81 | 98 | 28
  B/Florida [POST] | 106 | 114 | 31

10. Secondary Outcome: Number of Subjects Seroprotected Against HI Antibodies
Description: A seroprotected subject was defined as a vaccinated subject with serum HI titer ≥ 1:40.
  The flu strains assessed were the A/Brisbane (H1N1), A/Uruguay (H3N2) and B/Florida.
Time Frame: At Day 0 [PRE] and at Day 28 (for primed subjects) and at Day 56 (for unprimed subjects) [POST]
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Fluviral F1 Group | Fluviral F2 Group | Vaxigrip Group
Number analyzed (Participants) | 131 | 132 | 36
Participants
  A/Brisbane (H1N1) [PRE] | 17 | 21 | 5
  A/Brisbane (H1N1) [POST] | 70 | 84 | 30
  A/Uruguay (H3N2) [PRE] | 10 | 23 | 3
  A/Uruguay (H3N2) [POST] | 82 | 99 | 30
  B/Florida [PRE] | 17 | 20 | 7
  B/Florida [POST] | 111 | 122 | 33

11. Secondary Outcome: Seroconversion Factor for HI Antibodies
Description: The seroconversion factor (SCF) was defined as the fold increase in serum HI geometric mean titers (GMTs) post-vaccination (at Day 28 for primed subjects and at Day 56 for unprimed subjects) compared to pre-vaccination (Day 0).
  The flu strains assessed were the A/Brisbane (H1N1), A/Uruguay (H3N2) and B/Florida.
Time Frame: At Day 28 (for primed subjects) and at Day 56 (for unprimed subjects) [POST]
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | Fluviral F1 Group | Fluviral F2 Group | Vaxigrip Group
Number analyzed (Participants) | 131 | 132 | 36
fold increase
  A/Brisbane (H1N1) [POST] | 6.8 [5.2 to 8.9] | 8.3 [6.6 to 10.6] | 14.9 [9.6 to 23.3]
  A/Uruguay (H3N2) [POST] | 9.2 [7.3 to 11.7] | 9.7 [8.0 to 11.9] | 13.3 [8.9 to 19.9]
  B/Florida [POST] | 16.2 [12.8 to 20.5] | 20.7 [16.3 to 26.2] | 17.6 [10.4 to 29.9]

12. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms After Vaccination
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any solicited local symptom reported regardless of intensity grade. Grade 3 pain = Cried when limb was moved/spontaneously painful. Grade 3 redness and swelling were defined as redness/swelling above 50 millimeters (mm).
  This secondary outcome measure was assessed for the Vaxigrip Group as per the study protocol.
Time Frame: During the 4-day follow-up period (Days 0-3) after any vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaxigrip Group
Number analyzed (Participants) | 43
Participants
  Any pain | 17
  Grade 3 pain | 0
  Any redness | 13
  Grade 3 redness | 0
  Any swelling | 5
  Grade 3 swelling | 0

13. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms After Vaccination
Description: Symptoms assessed were drowsiness, irritability, loss of appetite and fever. Any was defined as occurrence of any general symptom regardless of their intensity grade or relationship to vaccination. Any fever = Axillary temperature ≥ 38.0 degrees Celsius (°C). Grade 3 fever = Axillary temperature ≥ 39.0°C. For other symptoms, grade 3 was defined as an adverse event which prevented normal everyday activities. Related = A general symptom assessed by the investigator as causally related to vaccination.
  This secondary outcome measure was assessed for the Vaxigrip Group as per the study protocol.
Time Frame: During the 4-day follow-up period (Days 0-3) after any vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaxigrip Group
Number analyzed (Participants) | 43
Participants
  Any drowsiness | 16
  Grade 3 drowsiness | 0
  Related drowsiness | 11
  Any irritability | 22
  Grade 3 irritability | 1
  Related irritability | 15
  Any loss of appetite | 14
  Grade 3 loss of appetite | 0
  Related loss of appetite | 9
  Any fever | 3
  Grade 3 fever | 0
  Related fever | 2

14. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs) After Vaccination
Description: Unsolicited AEs covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = Occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Grade 3 = Occurrence of any unsolicited AE that prevented normal, everyday activities. Related = Occurrence of an unsolicited AE assessed by the investigator to be causally related to study vaccination.
  This secondary outcome measure was assessed for the Vaxigrip Group as per the study protocol.
Time Frame: During the 28-day follow-up period (Days 0-27) after vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vaxigrip Group
Number analyzed (Participants) | 43
Participants
  Any unsolicited AE(s) | 24
  Grade 3 unsolicited AE(s) | 3
  Related unsolicited AE(s) | 8

15. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Medically-attended Adverse Events (MAEs) After Vaccination
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any MAE(s) = Occurrence of any MAE(s) regardless of intensity grade or relation to vaccination.
  Analysis of intensity and relationship to vaccination of MAEs was not performed.
  This secondary outcome measure was assessed for the Vaxigrip Group as per the study protocol.
Time Frame: During the 28-day post-vaccination period after vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vaxigrip Group
Number analyzed (Participants) | 43
Participants | 9

16. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Medically-attended Adverse Events (MAEs) After Vaccination
Description: as for outcome 15
Time Frame: During the 6-month safety follow up after vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vaxigrip Group
Number analyzed (Participants) | 43
Participants | 14

17. Secondary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs) After Vaccination
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any SAE(s) = Occurrence of any SAE(s) regardless of intensity grade or relation to vaccination. Related SAE(s) = Occurrence of any SAE(s) assessed by the investigator as causally related to vaccination.
  This secondary outcome measure was assessed for the Vaxigrip Group as per the study protocol.
Time Frame: During the 28-day post-vaccination period
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vaxigrip Group
Number analyzed (Participants) | 43
Participants
  Any SAE(s) | 0
  Related SAE(s) | 0

18. Secondary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs) After Vaccination
Description: as for outcome 17
Time Frame: During the 6-month safety follow up after vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vaxigrip Group
Number analyzed (Participants) | 43
Participants
  Any SAE(s) | 0
  Related SAE(s) | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed during the 28 day post vaccination period and the 6-month safety follow-up period. Systematically and non-systematically assessed frequent adverse events were assessed during 4 day and 28 day post vaccination periods.
Description: For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated cohort who had the symptom sheet completed. No related SAEs were reported.
Arm/Group | Fluviral F1 Group | Fluviral F2 Group | Vaxigrip Group
Serious Adverse Events (participants affected / at risk) | 2/164 | 2/167 | 0/43
Other Adverse Events (participants affected / at risk) | 129/164 | 138/167 | 34/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluviral F1 Group (N=164) | Fluviral F2 Group (N=167) | Vaxigrip Group (N=43)
Pneumonia (Infections and infestations) | 1 | 0 | 0 — SAE was assessed within the 28-day post vaccination period.
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — SAE was assessed within the 28-day post vaccination period.
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 — SAE was assessed through the 6-month safety follow-up period.
Viral pharyngitis (Infections and infestations) | 0 | 1 | 0 — SAE was assessed through the 6-month safety follow-up period.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Fluviral F1 Group (N=164) | Fluviral F2 Group (N=167) | Vaxigrip Group (N=43)
Pain (General disorders) | 45/161 | 55/164 | 17
Redness (General disorders) | 49/161 | 54/164 | 13
Swelling (General disorders) | 22/161 | 24/164 | 5
Drowsiness (General disorders) | 54/161 | 65/163 | 16
Irritability (General disorders) | 81/161 | 83/163 | 22
Loss of appetite (General disorders) | 50/161 | 54/163 | 14
Fever (General disorders) | 16/161 | 9/163 | 3
Diarrhoea (Gastrointestinal disorders) | 8 | 9 | 6
Teething (Gastrointestinal disorders) | 11 | 10 | 4
Vomiting (Gastrointestinal disorders) | 13 | 16 | 3
Pyrexia (General disorders) | 19 | 15 | 5
Nasopharyngitis (Infections and infestations) | 14 | 18 | 4
Upper respiratory tract infection (Infections and infestations) | 29 | 16 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 24 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.